CLINICAL TRIAL: NCT03144817
Title: Dialysate Sodium Lowering Trial
Acronym: DeSaLT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Dialysis Clinic, Inc. (Industry); InBody (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12393
Record Dates: First submitted 2017-04-27; First posted 2017-05-09 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Hemodialysis Complication; Fluid Overload; Dialysis Disequilibrium; Intra-dialytic Hypotension; Hypertension
Keywords: hemodialysis; fluid overload; dialysis disequilibrium; intra-dialytic hypotension; dialysate sodium lowering
MeSH Terms: conditions — Edema; Dysequilibrium syndrome; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental): Intervention group will dialyze with dialysate Na 135 mEq/L.
  Interventions: Other: Dialysate Sodium Lowering

INTERVENTIONS:
Other: Dialysate Sodium Lowering — Dialysate sodium is lowered until nadir sodium level is reached. Participant dialyzes at this sodium level until end of follow-up.
  Arms: Intervention Group

SUMMARY:
This is a pilot randomized clinical trial in which patients treated with 3X per weekly conventional hemodialysis will be treated to a dialysate sodium 135 mEq/L vs. 138 mEq/L and followed for safety and tolerability, effects on BP and volume.

DETAILED DESCRIPTION:
This is a pilot randomized clinical trial in which hypertensive hemodialysis patients will be randomized to a low dialysate sodium (Na) of 135 mEq/L or a standard dialysate Na of 138 mEq/L. Patients will be randomized 2:1 to the low arm. Dialysate Na will be lowered 1 mEq/L every 2 weeks, as tolerated. Tolerance will be assessed by symptoms, intradialytic hypotension (IDH) episodes (systolic BP <90 or intervention for symptoms or BP drop during dialysis), achievement of dry weight. The trial will last for 6 to 12 months, for an individual, depending on when they entered the trial. The primary outcome is feasibility and safety of using the lower dialysate sodium which is assessed by symptoms during or immediately after dialysis, intradialytic hypotension episodes and the frequency of emergency room visits and hospitalizations. Several secondary outcomes will be measured including blood pressure prior to dialysis and at home, change in plasma Na over time, dry weight, post-dialysis weight, interdialytic weight change, symptoms of thirst and dry mouth, self-reported dialysis recovery time, relative blood volume change during a single treatment (via 'Critline') and, in patients without an implanted electronic device, extraceullular fluid volume (via bioimpedance).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients undergoing thrice weekly in-center conventional HD
* At least 90 days since start of hemodialysis
* Absence of pulmonary edema / signs of fluid overload on physical exam
* Currently dialyzing at a DNa >=137 mEq/L
* Single session Kt/V >=1.3 each month for the past 2 months
* Hypertensive, defined by a pre-dialysis BP of >140/90 or treatment with 1 or more antihypertensive agents
* No more than 1 skipped treatment and no more than 1 session per month shortened by >10 min
* Life expectancy >12 months
* Able to provide Informed Consent
* Speaks and understands English

Exclusion Criteria:

* Prone to IDH, defined as IDH occurring in >10% of treatments in the past 3 months. IDH will be defined as symptoms (e.g. cramps, dizziness, loss of consciousness) and/or intra- or post-dialytic systolic BP <90 mm Hg and/or use of intervention(s) (UF goal lowered, treatment stopped early, or saline given) because of IDH
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Frequency of Intradialytic Hypotension | Baseline period through study completion, an average of 6 months
  IDH is determined by review of blood pressures (measured every 30 minutes during dialysis), symptoms (recorded by the nurse during the dialysis treatment and reviewed at Q2 weekly face to face visits by the study team) and the need for intervention (targeted ultrafiltration goal was reduced; treatment was terminated early or saline given for intradialytic hypotension. IDH is defined by any 1 (or more of the following) 1) lowest intradialytic Systolic BP <90 mm Hg or 2) intradialytic symptoms (cramps, lightheadedness, nausea +/-vomiting, diaphoresis, loss of consciousness or seizure) OR 3) intervention performed for symptoms of IDH or lowest intradialytic BP <90 mm Hg.
  The # IDH events (meeting 1 or more of the 3 criteria above) per 100 treatments will be compared across treatment arms.
Dialysis Dysequilibrium (Safety) | Baseline period through study completion, an average of 6 months
  Ascertained via self-report on a questionnaire that asks about the frequency of symptoms suggestive of DD occurring during or immediately after dialysis. The symptoms are: headache, nausea +/- vomiting, confusion, drowsiness, muscle twitching, blurred vision. There are 5 response options ranging from never through to very often for each question. The questionnaire is administered at baseline, at 6 weeks, and Q3 months thereafter. The change in frequency of each symptom will be compared across arms.
Frequency of ER visits and hospitalizations (safety) | Baseline through study completion
  The frequency of ER visits and hospitalizations will be ascertained at Q2 weekly study visits. The # of events per time at risk will be compared across treatment arms.
Frequency of patients treated to a dialysate Na 135 mEq/L at end of study (feasibility) | Last 2 weeks of Follow-up
  Among those assigned to Dialysate Na 135 mEq/l as the denominator, the # actually continuing to dialyze at this level during the last two weeks of study follow-up.

SECONDARY OUTCOMES:
Pre- and post-dialysis Plasma Sodium | Baseline period through study completion, an average of 6 months
  Taken from lab draws immediately before and after start of dialysis treatment.
Dialysate Sodium | Baseline period through study completion, an average of 6 months
  Sample of dialysate sodium taken 30 minutes after start of dialysis treatment.
Relative Blood Volume | Baseline period through study completion, an average of 6 months
  Determined using CRIT LINE III monitors.
Bioimpedance Analysis | Baseline period through study completion, an average of 6 months
  Water volume and bioimpedance results will be determined using InBodyS10 device.
Interdialytic Weight Gain | Baseline period through study completion, an average of 6 months
  Determined by analysis of treatment sheets.
Post Dialysis Weight | Baseline period through study completion, an average of 6 months
  Determined by analysis of treatment sheets.
Estimated Dry Weight | Baseline period through study completion, an average of 6 months
  Determined by analysis of treatment sheets.
Pre- and Post-dialysis Sitting Blood Pressure | Baseline period through study completion, an average of 6 months
  Determined by analysis of treatment sheets.
Home Blood Pressure Monitoring | Baseline period through study completion, an average of 6 months
  Participants will use a LifeSource blood pressure monitor to measure their blood pressure weekly at home.
Sodium Loss during Dialysis | Baseline period through study completion, an average of 6 months
  Calculated according to the formula: pre-dialysis total body Na - post-dialysis total body Na, where the volume of distribution in the extracellular space is estimated as 0.58*target weight.
Thirst and Xerostomia | Baseline through study completion, an average of 6 months
  Thirst and Xerostomia will be measured via validated, self-administered questionnaires, the 'Dialysis Thirst Inventory' and the 'Xerostomia Inventory' , respectively (BotsCP et al, Kidney International:66; 2004).
  Change in each inventory score from baseline to the end of the study will be compared by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Miskulin, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- DCI Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822